CLINICAL TRIAL: NCT06011694
Title: A Prospective, Multicenter Cohort Study of the Multi-omics Liquid Biopsy MCED Test MERCURY in an Average Risk Chinese Population
Brief Title: The Jinling Cohort
Status: Recruiting | Type: Observational
Sponsor: Nanjing Shihejiyin Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NanjingShihejiyinTech
Record Dates: First submitted 2023-08-09; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cancer; Multi Cancer Early Screening; Liquid Biopsy
Keywords: Early Detection of Cancer; MCED
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention: Each participant will undergo peripheral blood collection for MERCURY test, health questionnaires and annual routine physical exams once a year for three consecutive years, then followed up two additional years.
  Interventions: Other: MERCURY test, health questionnaires and annual routine physical exams

INTERVENTIONS:
Other: MERCURY test, health questionnaires and annual routine physical exams — Each participant will undergo peripheral blood collection for MERCURY test, health questionnaires and annual routine physical exams once a year for three consecutive years, then followed up two additional years.

SUMMARY:
The Jinling Cohort is a prospective, multicenter cohort study in which 15,000 eligible individuals aged 45-75 in Nanjing China will be enrolled.

DETAILED DESCRIPTION:
Its aim is to assess the performance and clinical utility of the Multi-omics liquid biopsy MCED test MERCURY in an average risk Chinese population. Each participant will undergo peripheral blood collection for MERCURY test, health questionnaires and annual routine physical exams once a year for three consecutive years, then followed up two additional years. The entire assess time is 60 months.

The primary goals of the study is to evaluate sensitivity, specificity, positive/negative predictive value and other performance of MERCURY test.

The secondary goal of the study is (1) to evaluate how many cancer types the test MERCURY can detect and TOO accuracy; (2) With MCED test and routine physical exams being conducted in parallel for three years and following up for five years, the study allows to assess MERCURY test can detect cancer how many years earlier than conventional methods, leading to its clinical value evaluation of whether it can ensure reduction in late-stage cancer diagnosis; (3) to evaluate participants' attitude and perception towards MCED blood test.

ELIGIBILITY:
Inclusion Criteria:

1、45-75 years of age; 2、Willing and able to undergo blood sample collection, health questionnaires and annual routine physical exams once a year for three consecutive years; 3、Residents in Nanjing; 4、Fully understand the study and able to provide a written informed consent

Exclusion Criteria:

1. Pregnant women;
2. Individuals who have history of cancer or current diagnosis of cancer;
3. Individuals who have organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant;
4. Individulas who have blood transfusion within 30 days prior to the blood draw;
5. Individuals who have an acute infection or inflammation within 14 days prior to the blood draw;
6. Individuals who have taken medication with anti-tumor effects within 30 days prior to the blood draw;
7. Individuals who will not be able to comply with the protocol procedures judged by researchers

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 45 Years to 75 Years (Adult, Older Adult)，Each participant will undergo peripheral blood collection for MERCURY test, health questionnaires and annual routine physical exams once a year for three consecutive years, then followed up two additional years.
  No
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate sensitivity, specificity, positive/negative predictive value and other performance measures of the multi-omics liquid biopsy test MERCURY for multi-cancer early detection in average risk population | assessed up to 60 months

SECONDARY OUTCOMES:
To evaluate how many cancer types the multi-omics liquid biopsy MCED (multi-cancer early detection) test MERCURY can detect and TOO (tumor of origin) accuracy | assessed up to 60 months
  To assess whether the TOO (tumor of origin) results predicted from the multi-omics liquid biopsy MCED (multi-cancer early detection) test MERCURY match with clinical diagnostic tumor types received from follow-up. Summarize the number of consistency and inconsistency to evaluate the prediction accuracy
To assess test MERCURY's efficiency and clinical utility in average risk population | assessed up to 60 months
  To assess MERCURY test's lead-time relative to clinical diagnosis. With MCED test and routine physical exams being conducted in parallel for three years and following up for five years, the study allows to assess MERCURY test can detect cancer how many years earlier than conventional methods by comparing MERCURY test positive timepoint to tumor clinical diagnosis timepoint.
To evaluate participants' attitude and perception towards MCED blood test | assessed up to 60 months
  To compare the adherence to annual blood exams to reported SOC (standard of care) screening methods to see whether participants' perception towards MCED blood test

CONTACTS AND LOCATIONS:
Overall Officials: Shao Yang, Ph.D, Principal Investigator — NanjingShihejiyin Technology Inc.
Locations (2):
- China (2):
  - Nanjing Jiangbei People's Hospital, Nanjing, Jiangsu
  - The Fourth Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No